CLINICAL TRIAL: NCT04070443
Title: A Multicentre, Open-label Phase II Trial Evaluating the Safety and Efficacy of Ponatinib Induction Followed by Imatinib Maintenance in Adult Patients With Chronic Myelogenous Leukemia in Chronic Phase (CML-CP) ≤ 65 Years
Brief Title: Safety and Efficacy of Ponatinib Followed by Imatinib in Patients With Chronic Myelogenous Leukemia in Chronic Phase
Acronym: TIPI
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ET18000120 (TIPI)
Record Dates: First submitted 2019-07-19; First posted 2019-08-28 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Philadelphia Chromosome Positive CML; BCR-ABL Positive Chronic Myelogenous Leukemia
Keywords: Clinical Trial, Phase II; Tyrosine Kinase Inhibitors; Induction phase; Consolidation phase
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — ponatinib; Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Induction phase with Ponatinib followed by Imatinib (Experimental): Ponatinib (Iclusig®) : Tyrosine Kinase Inhibitor (BCR-ABL); oral (tablets) : 30mg/day during 6 months (induction phase); Takeda & Incyte Biosciences.
  Imatinib (either Glivec® or any generic form) : Tyrosine Kinase Inhibitor (BCR-ABL, ABL, KIT and PDGFRA receptor tyrosine kinases); oral : 400 mg/day during at least 30 months (then, depending of MR4.5)
  Interventions: Drug: Ponatinib; Drug: Imatinib

INTERVENTIONS:
Drug: Ponatinib — 30mg/day; 6 months. Dose adaptation procedures are planned in case of toxicity.
Drug: Imatinib — 400 mg/day; at least 30 months (M7 to M36), then depending of MR4.5 . Dose adaptation procedures are planned in case of toxicity.

SUMMARY:
The investigators hypothesize that, in newly diagnosed de novo chronic phase CML patients, an induction treatment with ponatinib for 6 months should increase the rate of patients reaching a stable MR4.5 allowing cessation of imatinib treatment.

The investigators proposal is to conduct a multicenter, Phase II trial to evaluate the safety, clinical and biological activity of an induction treatment with ponatinib for 6 months, followed by a consolidation treatment with imatinib in newly diagnosed de novo chronic phase CML patients.

DETAILED DESCRIPTION:
TREATMENT PLAN :

All eligible patients will be treated:

* During the induction Phase (Month 1 to Month 6) with ponatinib (30mg/day) single agent; then
* During the consolidation Phase (Month 7 to Month 36) with imatinib (400mg/day) single agent; then
* From M36 :

  * Patients with stable MR4.5 (i.e. since at least 2 years) will enter in the TFR phase and will stop imatinib treatment. Thereafter, in case of MMR loss, imatinib will be re-introduced as per investigator judgement (including for dose).
  * Patients without stable MR4.5 will continue imatinib treatment until stable MR4.5, or M60, PD, death, withdrawal of consent or overall trial completion. Such patients will be allowed to enter into the TFR phase as soon as a stable 2-year MR4.5 is reached: however, they will be considered as a failure for the primary endpoint analysis.

STATISTICS :

A total of 170 patients will be enrolled in this study.

According to a Fleming design, with a P0=20% as minimal efficacy rate and P1=30% as an expected target, 156 patients should be enrolled, assuming an unilateral type I error alpha of 5% and 90% power. At the time of analysis, if at least 40 successes are observed among the 156 evaluable patients, the treatment will be considered as interesting for further investigation in this indication. Considering that some patients may withdraw their consent before 36 months (about 10%), the investigators plan to enrol 170 patients in total.

DATA ENTRY, DATA MANAGEMENT AND STUDY MONITORING All the data concerning the patients will be recorded in the electronic case report form (eCRF) throughout the study. Serious adverse event (SAE) and Adverse Event of Specific Interest (AESI) reporting will be also paper-based by e-mail and/or Fax.

The sponsor will perform the study monitoring and will help the investigators to conduct the study in compliance with the clinical trial protocol, Good Clinical Practices (GCP) and local law requirements.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged ≥18 and ≤65 years at time of inform consent signature.
* Cytologically confirmed CML, Philadelphia chromosome positive with or without additional chromosomal abnormalities and/or BCR-ABL positive (Major BCR (M-BCR) transcript exclusively), i. e. Cryptic Philadelphia chromosome patients can be enrolled:

  * diagnosed within the past 3 months prior to D1 (i.e. within 60 days [± 7 days] since the date of first cytogenetic analysis),
  * in chronic phase defined by i) <15 % blasts in peripheral blood and bone marrow, ii) < 30% blast plus promyelocytes in peripheral blood and bone marrow; iii) < 20 % basophils in peripheral blood and iv) ≥100 X 109 platelets/L in peripheral blood,
  * no extra-medullary disease.
  * All EUTOS long-term survival Scores.
* No prior treatment for CML with any tyrosine kinase inhibitor (eg. imatinib, dasatinib, nilotinib or bosutinib), or busulphan; interferon-alpha; homoharringtonine; cytosine arabinoside; or any other investigational agent; with the exception of hydroxyurea and/or anagrelide which are the only authorized prior treatments.

Note: Hydroxyurea should be stopped at least 24 hours prior the initiation of ponatinib.

* Eastern Cooperative Oncology Group performance status (ECOG PS) of 0, 1 or 2.
* Adequate organ functions as defined below according to lab tests performed within 7 days before Day 1:

Renal function:

- Serum creatinine clearance ≥ 50 mL/min/1.73m2 according to CKD-EPDI formula or serum creatinine ≤ 2 upper limit of normal (ULN).

Hepatic function:

* Serum bilirubin < 1.5 × ULN, with the following exception: Patients with known Gilbert disease who have serum bilirubin level ≤ 3 ULN may be enrolled.
* Aspartate aminotransferase (AST), alanine aminotransferase (ALT) and alkaline phosphatase ≤ 2.5 ULN.
* Amylase or Lipase ≤ 1.5 × ULN Total cholesterol ≤1.5 ULN

  * Women of child-bearing potential must have a negative serum pregnancy test within 7 days before study drug start and must agree to use an effective form of contraception from the time of the negative pregnancy test up to 3 months after the last dose of study treatments.
  * Fertile men must agree to use an effective method of contraception during the study and for up to 3 months after the last dose of study treatments.
  * Patient should understand, sign, and date the written voluntary informed consent form prior to any protocol-specific procedures performed. Patient should be able and willing to comply with study visits and procedures as per protocol.
  * Patients must be covered by a medical insurance.

Exclusion Criteria:

* Any form of prior auto- or allo-hemopoietic stem cell transplant.
* Hypersensitivity to the active substance or to any of the excipients of ponatinib and imatinib (see respective IB/SmPC).
* Inability to take oral medication including malabsorption syndrome or other illness that could affect oral absorption of the study treatments (hereditary problems of galactose intolerance, the Lapp lactase deficiency or glucose-galactose malabsorption).
* Patients using, or requiring to use while on the study of any not permitted concomitant medications:

  * Any approved anti-cancer systemic treatment including chemotherapy, targeted therapy, immunotherapy or any biological therapy,
  * Any investigational agents,
  * Any treatment able to induce " torsades de pointes ",
  * Any strong inducers and inhibitors of CYP3A4.
* Patients with a malignancy other than CP-CML within 5 years prior to Day 1 with the exception of those with a negligible risk of metastasis or death and treated with expected curative outcome (such as adequately treated in situ carcinoma of the cervix, basal or squamous cell skin cancer, localised prostate cancer or ductal in situ carcinoma treated surgically with curative intent).
* Patients with active B or C hepatitis infection. Notes: Patients with past Hepatitis B Virus (HBV) infection or resolved HBV infection (defined as having a negative hepatitis B surface antigen (HBsAg) test and a positive hepatitis B core antibody (HBcAb) test) are eligible.

Patients with a positive HBcAb test must have a negative HBV DNA test at screening.

Patients positive for Hepatitis C Virus (HCV) antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV RNA.

* Patients with significant cardiovascular disease, such as New York Heart Association cardiac disease Class II or greater, myocardial infarction within 3 months prior to D1, unstable arrhythmias, unstable angina, peripheral arterial occlusive disease, venous thromboembolism or pulmonary embolism, brain stroke, evolutive ischemic cardiopathy; prolonged corrected QT interval (QTc) interval on baseline electrocardiogram (>450 msec on the Fridericia's correction) despite correction of predisposants factors; long congenital QT syndrome.
* Any of the following medical conditions despite adequate therapeutic management:

  * Uncontrolled HTA despite adequate ongoing treatment.
  * Diabetes with documented target organ damage.
* Pregnant or lactating women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2019-11-13 (Actual); Primary Completion 2029-06-01 (Estimated); Study Completion 2029-06-01 (Estimated)

PRIMARY OUTCOMES:
Impact of Ponatinib induction treatment on the TFR rate | 36 months after initiation of ponatinib
  Rate of patients reaching a stable MR4.5 (BCR-ABL (IS) ≤0.0032% with at least 32,000 copies of ABL) for ≥ 2 years from Month 36 after initiation of ponatinib.

SECONDARY OUTCOMES:
Clinical activity of the proposed therapeutic strategy | up to 24 months after ponatinib initiation
  For all patients : Rate of patients with MR4.5; MR4.0 and MMR at 1, 2, 3, 6, 9, 12, 24 months after ponatinib initiation
Clinical activity of the proposed therapeutic strategy | up to 6 months after ponatinib initiation
  For all patients : Rate of patients with a BCR-ABL/ABL (IS) ≤ 10% and rate of patients with CCyR (or its molecular equivalent, BCR-ABL/ABL (IS) ≤ 10%) at 3 and 6 months after ponatinib initiation.
Clinical activity of the proposed therapeutic strategy | from the first intake of Ponatinib until one of this criteria is reached, assessed up to 5 years
  For all patients : Time to MR4.5, MR4.0 or MMR following ponatinib initiation
Clinical activity of the proposed therapeutic strategy | from the first intake of Ponatinib until one of this criteria is reached, assessed up to 5 years
  For all patients : Duration of MR4.5, MR4.0 or MMR
Clinical activity of the proposed therapeutic strategy | from the date of inclusion until the date of the first progression or date of death from any cause, whichever came first, assessed up to 5 years
  For all patients : Progression Free survival
Clinical activity of the proposed therapeutic strategy | From the date of inclusion until the date of death from any cause, whichever came first, assessed up to 5 years
  For all patients : Overall survival
Clinical activity of the proposed therapeutic strategy | 3, 6, 9, 12 and 24 months after imatinib cessation
  For patients reaching TFR criteria and following imatinib cessation: Rate of successful TFR (patients sill with MR4.5) at 3, 6, 9, 12 and 24 months after imatinib cessation
Clinical activity of the proposed therapeutic strategy | from imatinib cessation until the date of progression/relapse, whichever came first, assessed up to 5 years
  For patients reaching TFR criteria and following imatinib cessation: Duration of TFR after imatinib cessation.
Clinical activity of the proposed therapeutic strategy | From the date of imatinib cessation until the date of death from any cause, assessed up to 5 years
  For patients reaching TFR criteria and following imatinib cessation: OS after imatinib cessation
Clinical activity of the proposed therapeutic strategy | from the date of imatinib cessation until the date of the first progression or date of death from any cause, whichever came first, assessed up to 5 years
  For patients reaching TFR criteria and following imatinib cessation: PFS after imatinib cessation
Clinical activity of the proposed therapeutic strategy | from the date of ponatinib initiation until the onset of the following events: loss of responses, accelerated phase or blast crisis at any time, death at any time from any cause; drug discontinuation due to adverse events, assessed up to 5 years
  For patients reaching TFR criteria and following imatinib cessation: Event-free survival according ELN recommendations
Clinical activity of the proposed therapeutic strategy | from the date of imatinib cessation until 30 days after the last study drugs intake or until initiation of a new anti-cancer treatment, whichever came first, assessed up to 5 years
  For patients reaching TFR criteria and following imatinib cessation: Rate of TKI-withdrawal syndrome after Imatinib cessation
Clinical activity of the proposed therapeutic strategy | from the date of imatinib re introduction until date of MMR or MR4.5, assessed up to 5 years
  For patients reaching TFR criteria and following imatinib cessation: Rate of MMR, MR4.0 and MR4.5 recovery in case of imatinib re-introduction (
Incidence of Adverse Events of the proposed therapeutic strategy | from the signature of the ICF and the first intake of study drug until 30 days after the last study drugs intake or until initiation of a new anti-cancer treatment, assessed up to 5 years
  * Hematologic and non-hematologic AEs graded according to the NCI CTCAE v5.0
  * Incidence of arterial thrombotic events during the induction phase and during the consolidation phase.
Quality of Life (QLQ-CML24 questionnaire) | At screening, at each visit from Month 1 to Month 60 (if applicable) and then during the TFR phase and at STSV 30 days, assessed up to 5 years
  Evolution of Quality of life according to QLQ-CML24 questionnaire.
Quality of Life (QLQ-C30 questionnaire) | At screening, at each visit from Month 1 to Month 60 (if applicable) and then during the TFR phase and at STSV 30 days, assessed up to 5 years
  Evolution of Quality of life according to QLQ-C30 questionnaire.
Ponatinib pharmacokinetics (non-decisional) | At screening, at each visit from Month 6 (induction phase)
  Plasma concentrations of ponatinib over the 6 months of the induction period.
Patient' compliance to the proposed therapeutic strategy | At each visit during induction and consolidation phase
  Compliance to ponatinib and imatinib as evaluated using the Morisky medication adherence scale questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Franck-Emmanuel NICOLINI, MD, Principal Investigator — Centre Leon Berard
Locations (28):
- France (28):
  - Chu Amiens Picardie, Amiens
  - CHU d'Angers, Angers
  - Centre Hospitalier Annecy-Genevois, Annecy
  - CH d'Avignon, Avignon
  - Chru Besançon, Besançon
  - Institut Bergonie, Bordeaux
  - Chru Brest, Brest
  - Institut D'Hematologie de Basse Normandie, Caen
  - Chu D'Estaing, Clermont-Ferrand
  - Centre Hospitalier Sud Francilien, Corbeil-Essonnes
  - Hopital Henri Mondor, Créteil
  - CHU de Grenoble, Grenoble
  - CH de Versailles - Hôpital André Mignot, Le Chesnay
  - Hôpital Claude Huriez - CHRU de Lille, Lille
  - CHU Limoges - Hôpital Dupuytren, Limoges
  - Centre Léon Bérard, Lyon
  - Institut Paoli Calmettes, Marseille
  - Hopital Saint Eloi, Montpellier
  - Chu Hotel Dieu, Nantes
  - CHU Nîmes Caremeau - Institut de Cancérologie du Gard, Nîmes
  - Hopital Saintantoine, Paris
  - Chu Poitiers, Poitiers
  - Chu - Hopital de Pontchaillou, Rennes
  - Institut de Cancérologie Lucien Neuwirth, Saint-Priest-en-Jarez
  - CHU Strasbourg, Strasbourg
  - Iuct Toulouse - Oncopole, Toulouse
  - CHRU Nancy/Brabois, Vandœuvre-lès-Nancy
  - Hopital Paul Brousse, Villejuif

IPD SHARING:
Plan to Share IPD: No